CLINICAL TRIAL: NCT03192254
Title: Understanding Mechanisms of Health Behavior Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Angela Bryan, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-0700
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obesity; Diet Modification; Incentives
MeSH Terms: conditions — Overweight; Obesity | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Monitoring Control (Active Comparator): Daily tracking of fruit and vegetable consumption
  Interventions: Behavioral: self-monitoring
- Daily Incentives (Experimental): Incentives for fruit and vegetable consumption delivered daily
  Interventions: Behavioral: self-monitoring; Behavioral: daily monetary incentives
- Delayed Lump Sum Incentives (Experimental): Incentives for fruit and vegetable consumption delivered in a lump sum at the end of the intervention
  Interventions: Behavioral: self-monitoring; Behavioral: delayed lump sum monetary incentives

INTERVENTIONS:
Behavioral: self-monitoring — recording fruit and vegetable consumption
Behavioral: daily monetary incentives — daily payments for consuming fruits and vegetables
  Arms: Daily Incentives
Behavioral: delayed lump sum monetary incentives — lump sum payments for consuming fruits and vegetables
  Arms: Delayed Lump Sum Incentives

SUMMARY:
This research seeks to examine psychological factors that may impact relationship between incentives and health behavior engagement, specifically fruit and vegetable consumption. Additionally, it will compare the impact of two different incentive schedules on behavior engagement, one providing immediate rewards (i.e. rewards received on a daily basis) and another providing delayed rewards (i.e. rewards received at the end of the study period), with a control condition in which no rewards are offered. Study participants will provide reports of their fruit and vegetable consumption each day for three weeks, and in the two incentive conditions, they will receive small monetary rewards for their fruit and vegetable consumption. Following the three week reporting and reward period, participants will complete two additional assessments, measuring psychological constructs and behavior engagement following the cessation of rewards. The study will also examine how cognitive and anthropomorphic factors may contribute to intervention response and the effects on psychological constructs.

ELIGIBILITY:
Inclusion Criteria:

* Consume fewer than 3 servings/day of fruits and vegetables
* Daily access to internet for 3 weeks following baseline session
* Have or are willing to create an account on PayPal
* BMI greater than or equal to 25, from self-reported height and weight

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable consumption, servings per week | 3 Weeks
Fruit and vegetable consumption, servings per week | 5 Weeks
Perceived behavioral control scale score | 3 Weeks
Perceived behavioral control scale score | 5 Weeks
Attitude scale score | 3 Weeks
Attitude scale score | 5 Weeks

SECONDARY OUTCOMES:
Intrinsic motivation scale score | 3 Weeks
Intrinsic motivation scale score | 5 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No